CLINICAL TRIAL: NCT02159079
Title: A Phase II/III Randomized Controlled Trial of a Conservative Fluid Balance Strategy for Patients With Sepsis and Cardiopulmonary Dysfunction
Brief Title: A Randomized Controlled Trial of a Conservative Fluid Balance Strategy for Patients With Sepsis and Cardiopulmonary Dysfunction (BALANCE Study)
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Matthew Semler, Fellow in Pulmonary and Critical Care Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140582
Record Dates: First submitted 2014-06-03; First posted 2014-06-09 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Sepsis
Keywords: Sepsis; Severe Sepsis; Septic Shock; Conservative Fluid Management; Fluid Balance; Fluid Restriction
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Patients in the usual care arm will be managed exclusively by their treating clinician without input from study personnel.
- Conservative Fluid Management Strategy (Experimental): For patients in the conservative fluid management arm, beginning 12 hours after admission to study ICU and ending at the first of ICU discharge, death, return to home inspired oxygen, or study day 14, fluid management will be controlled by a study protocol. Patients in shock will receive fluid boluses only as specified by the protocol for oliguria and rapidly increasing vasopressor requirement. Patients not in shock will receive fluid boluses only as specified by the protocol for oliguria. Output will exceed input each day using a diuretic drip if required. Study protocol will be held only for pre-specified Safety Endpoints of persistent oliguria, decompensating shock, diuretic side effect, and intervening acute event.
  Interventions: Other: Conservative Fluid Management Strategy

INTERVENTIONS:
Other: Conservative Fluid Management Strategy — For patients in the conservative fluid management arm, beginning 12 hours after admission to study ICU and ending at the first of ICU discharge, death, return to home inspired oxygen, or study day 14, fluid management will be controlled by a study protocol. Patients in shock will receive fluid boluses only as specified by the protocol for oliguria and rapidly increasing vasopressor requirement. Patients not in shock will receive fluid boluses only as specified by the protocol for oliguria. Output will exceed input each day using a diuretic drip if required. Study protocol will be held only for pre-specified Safety Endpoints of persistent oliguria, decompensating shock, diuretic side effect, and intervening acute event.
  Arms: Conservative Fluid Management Strategy

SUMMARY:
Sepsis is a common inflammatory response to infection characterized by hypovolemia and vasodilation for which early administration of intravenous fluids has been suggested to improve outcomes. The ideal fluid balance following initial resuscitation is unclear. Septic patients treated in the intensive care unit commonly receive significant volumes of intravenous fluids with resultant positive fluid balance for up to a week after their initial resuscitation. Observational studies have associated fluid receipt and positive fluid balance in patients with severe sepsis and septic shock with increased mortality but are inherently limited by indication bias. In order to determine the optimal approach to fluid management following resuscitation in patients with severe sepsis and septic shock, a randomized controlled trial is needed. The primary hypothesis of this study is that, compared to usual care, a conservative approach to fluid management after resuscitation in patients with sepsis and cardiopulmonary dysfunction will increase intensive care unit free days.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients
* Adults
* Sepsis as defined by at least two systemic inflammatory response syndrome criteria and receipt of antimicrobial therapy
* Cardiopulmonary dysfunction as defined shock or respiratory failure

Exclusion Criteria:

* Inability to obtain consent
* Greater than 48 hours since inclusion criteria initially met
* Allergy to furosemide AND bumetanide
* Rhabdomyolysis with creatinine kinase > 5000 U/L
* Hypercalcemia with calcium >11 mg/dL
* Diabetic Ketoacidosis requiring continuous insulin infusion
* Tumor Lysis Syndrome diagnosed clinically
* Pancreatitis diagnosed clinically
* Chronic Hypoxic Respiratory Failure with Home Oxygen Use of FiO2≥0.3
* Chronic ventilator dependence
* cervical spinal cord injury at level C5 or higher
* amyotrophic lateral sclerosis
* Guillain-Barré Syndrome
* myasthenia gravis
* Renal failure requiring renal replacement therapy
* Burns >20% of body surface area
* Pregnant
* Preexisting pulmonary hypertension with PAPmean>40 on RHC
* Severe chronic liver disease with Childs-Pugh Score >11
* Moribund and not expected to survive an additional 24 hours
* Actively withdrawing life support or transitioning to comfort measures only
* Unwillingness of treating physician to employ conservative fluid strategy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W. Semler, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Semler MW, Janz DR, Casey JD, Self WH, Rice TW. Conservative Fluid Management After Sepsis Resuscitation: A Pilot Randomized Trial. J Intensive Care Med. 2020 Dec;35(12):1374-1382. doi: 10.1177/0885066618823183. Epub 2019 Jan 10. PMID 30630380

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Conservative Fluid Management Strategy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Conservative Fluid Management Strategy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [57 to 77] | 61 [54 to 75] | 63 [55 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: ICU-free Days to 14 Days After Enrollment
Description: The primary outcome will be the number of ICU-free days to day 14 (defined as the number days alive and outside of the intensive care unit in the first 14 days after enrollment).
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Conservative Fluid Management Strategy
Number analyzed (Participants) | 15 | 15
days | 9 [0 to 12] | 11 [0 to 12]

2. Secondary Outcome: Ventilator-free Days to Day 14
Description: A secondary outcome will be the number of ventilator-free days (defined as the number of days alive and breathing unassisted after the final achievement of unassisted breathing before day 14)
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Conservative Fluid Management Strategy
Number analyzed (Participants) | 15 | 15
days | 13 [0 to 14] | 12 [0 to 14]

3. Secondary Outcome: In-hospital Mortality to Day 14
Description: A secondary outcome will be in-hospital mortality to day 14 (defined as the incidence of mortality prior to hospital discharge within 14 days after enrollment).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Conservative Fluid Management Strategy
Number analyzed (Participants) | 15 | 15
Participants | 4 | 3

4. Secondary Outcome: Renal Replacement Therapy-free Days to Day 14
Description: Renal replacement therapy-free days to day 14 (defined as the number of days alive and free of renal replacement therapy from the last receipt of renal replacement therapy after enrollment to study day 14)
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Conservative Fluid Management Strategy
Number analyzed (Participants) | 15 | 15
days | 14 [0 to 14] | 14 [14 to 14]

5. Secondary Outcome: Highest Stage of Acute Kidney Injury
Description: Highest stage of acute kidney injury as defined according to Kidney Disease Improving Global Outcomes (KDIGO) criteria Stage 0 (no acute kidney injury) Stage 1 Serum creatinine 1.5-1.9 times baseline or ≥0.3 mg/dl (≥26.5 mmol/l) increase or Urine output <0.5 ml/kg/h for 6-12 hours Stage 2 Serum creatinine 2.0-2.9 times baseline or <0.5 ml/kg/h for ≥12 hours Stage 3 Serum creatinine 3.0 times baseline or Increase in serum creatinine to ≥4.0 mg/dl (≥353.6 mmol/l) or Initiation of renal replacement therapy or in patients <18 years, decrease in eGFR to <35 ml/min per 1.73 m² or Urine output <0.3 ml/kg/h for ≥24 hours or anuria for ≥12 hours
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Conservative Fluid Management Strategy
Number analyzed (Participants) | 15 | 14
Participants
  No acute kidney injury | 5 | 6
  Stage I | 0 | 2
  Stage II | 4 | 3
  Stage III | 6 | 3

6. Secondary Outcome: Highest Plasma Creatinine Between Enrollment and 28 Days After Enrollment
Description: Highest plasma creatinine (mg/dL) between enrollment and 28 days after enrollment, censored at hospital discharge
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Usual Care | Conservative Fluid Management Strategy
Number analyzed (Participants) | 15 | 15
mg/dL | 2.3 [1.1 to 3.1] | 1.3 [0.8 to 2.1]

7. Secondary Outcome: Receipt of Renal Replacement Therapy
Description: receipt of renal replacement therapy between enrollment and the first of 28 days or hospital discharge
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Conservative Fluid Management Strategy
Number analyzed (Participants) | 15 | 15
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 28 days
Description: Adverse event is defined as any untoward medical occurrence in a patient who participates in the study, without regard to a causal relationship. Death and organ dysfunction occur commonly in the ICU and are expected outcomes, therefore, for the purposes of this study, death and organ dysfunction will not be recorded as adverse events unless the investigator believes the event may have been caused by the study.
Arm/Group | Usual Care | Conservative Fluid Management Strategy
All-Cause Mortality (participants affected / at risk) | 4/15 | 3/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No